CLINICAL TRIAL: NCT02654431
Title: Identification and Semi -Quantification of ER/PR Proteins Expression Status in Formalin Fixed, Paraffin-embedded Normal and Neoplastic Tissue
Brief Title: Identification and Semi -Quantification of ER/PR Proteins Expression
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASI-ER/PR-IHC
Record Dates: First submitted 2014-06-26; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Immunohistochemical (IHC); ER/PR; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breast Cancer patients: Breast cancer patients
  Interventions: Procedure: Breast Cancer patient; Procedure: Cancer patients
- women with breast cancer: women with breast cancer
  Interventions: Procedure: Breast Cancer patient; Procedure: Cancer patients
- Cancer patients: Cancer patients
  Interventions: Procedure: Breast Cancer patient; Procedure: Cancer patients

INTERVENTIONS:
Procedure: Breast Cancer patient — Samples
Procedure: Cancer patients — Samples

SUMMARY:
The purpose of the study is the identification and quantification of proteins expression level in breast cancer tissues.

The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classifying ER/PR IHC stained samples.

DETAILED DESCRIPTION:
The anti ER/PR Kit is a semi-quantitative immunohistochemical (IHC) assay to identify the progesterone (PR) and estrogen (ER) expressions in formalin-fixed, paraffin-embedded human breast cancer tissue specimens. Results from the ER/PR test is indicated as an aid in the assessment of the hormones status of breast cancer patients. While the ER/PR kit provides the antibodies that offer direct visualization and semi-quantification of the protein expression through a brightfield microscope, the GenASIs GoPath system is designed to complement the routine workflow of the pathologist in the review of immunohistochemically stained histologic slides.

ELIGIBILITY:
Inclusion Criteria:

* Women having breast cancer

Exclusion Criteria:

* others

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
IVD study of ER/PR IHC samples: Accuracy of analysis | 1 Day
  Comparison tests (accuracy) between manual and automatic analysis of antibody expressions. The results from the automatic counting from the clinical studies will be compared to the manual counting analysis.
  Accuracy of the study will be declared "Success" if Positive, Negative and Overall agreement with manual count of the ER & PR antibody at least 90%.
IVD study of ER/PR IHC samples: Repeatability & Reproducibility of analysis | 1 Day
  Repeatability & Reproducibility tests of system analysis of antibody expressions. R&R acceptance criteria of ER/PR are related to the average agreement for between runs, between days and between systems R&R part of the study will be declared "Success" if Positive and Negative average agreement will be at least 85%.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Dobin, Study Chair — Section Chief, Cytogenetics
Locations (1):
- Scott & White Hospital,,, Temple, Texas, United States